CLINICAL TRIAL: NCT05893758
Title: A Real-world Registry Assessing the Clinical Use of the Lifetech Cera™ PFO Occluder
Brief Title: Lifetech Cera™ PFO Occluder Post-Market Clinical Follow-Up
Status: Completed | Type: Observational
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LT-TS-275-2023-02
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Patent Foramen Ovale; PFO
Keywords: Lifetech; Cera PFO; Occluder
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PFO subjects: Patients with a confirmed diagnosis of Patent Foramen Ovale (PFO) which is associated with TIA or cryptogenic stroke, and implanted with the investigational device.
  Interventions: Device: The Cera™ PFO Occluder

INTERVENTIONS:
Device: The Cera™ PFO Occluder — The Cera™ PFO Occluder is a percutaneous, transcatheter closure device for the non-surgical closure of Patent Foramen Ovale (PFO).

SUMMARY:
The objective of this post-market registry is to assess the clinical use of the Lifetech Cera™ PFO Occluder in a real-world and on-label fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of Patent Foramen Ovale (PFO);
2. Associated with TIA or cryptogenic stroke;
3. Patients was implanted with the investigational device as per IFU instructions;
4. Patients or legally authorized representatives have signed Data Release Consent or equivalent documents.

Exclusion Criteria:

1. Any contraindication mentioned in the corresponding IFU;
2. Patients did not conduct any follow up visit after hospital discharge.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of Patent Foramen Ovale (PFO) which is associated with TIA or cryptogenic stroke, and implanted with the investigational device.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of stroke/TIA, procedure/device-related death and serious procedure/device complications | from attempted procedure to 24 months post-implantation.
  Serious procedure/device complications include device embolization, cardiac or vascular perforation, atrial fibrillation, device thrombosis, pulmonary embolism and deep vein thrombosis.

SECONDARY OUTCOMES:
Successful closure of the PFO, confirmed by contrast Transcranial Doppler (cTCD), defined as with no, small or moderate residual shunt | at procedure, 6 months and 12 months post-implantation
Incidence of device or procedure related Adverse Events (AEs) | from attempted procedure to 24 months post-implantation
Incidence of device or procedure related Serious Adverse Events (SAEs) | from attempted procedure to 24 months post-implantation
Incidence of Device Deficiencies (DD) | from attempted procedure to 24 months post-implantation
Incidence of death | from attempted procedure to 24 months post-implantation

CONTACTS AND LOCATIONS:
Locations (5):
- Poland (5):
  - Oddział Kardiologii, Pracownia Hemodynamiki, Oddział Intensywnego Nadzoru Kardiologicznego oraz Pracownia Elektrofizjologii w Szpitalu w Myszkowie G.V.M.Carint, Myszków
  - Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii G.V.M.Carint-Oświęcim, Oświęcim
  - Polsko-Amerykańskie Kliniki Serca, Centrum Sercowo- Naczyniowe w Tychach, Grupa American Heart of Poland, Tychy
  - Polsko-Amerykańskie Kliniki Serca I Oddział Kardiologii Inwazyjnej i Niewydolności Serca w Ustroniu, Grupa AHoP, Ustroń
  - Szpital Powiatowy im. dr Tytusa Chałubińskiego w Zakopanem, Zakopane

IPD SHARING:
Plan to Share IPD: No